CLINICAL TRIAL: NCT06833242
Title: Single-plane Versus Real-time Biplane Approaches for Ultrasound-Guided Hip Joint Injection: A Prospective Randomized Controlled Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Mao (Other)
Responsible Party: Sponsor-Investigator, Yi Mao, clinician, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ChinaPLAGH20250213
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Hip Pain
Keywords: Hip Joint; Puncture; Injection; Single-plane; Real-time biplane

STUDY DESIGN:
Masking Description: There are practical differences in operation and blind methods cannot be achieved.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The real-time biplane ultrasound guidance group (Experimental): For the real-time biplane ultrasound guidance group, the hip joint injections was performed under the guidance of Xplane ultrasound with a X6-1 volume transducer probe (frequency range 1.0-6.0MHz).
  Interventions: Device: Real-time 3D Xplane ultrasound
- The single-plane ultrasound guidance group (No Intervention): For the single-plane ultrasound guidance group, the hip joint injections was performed under the guidance with a C5-1 convex array transducer (frequency range1.0-5.0 MHz)

INTERVENTIONS:
Device: Real-time 3D Xplane ultrasound — After the puncture needle is in the skin, the longitudinal section of the Xplane mode can be adjusted to keep the needle in the proposed plane.
  Arms: The real-time biplane ultrasound guidance group

SUMMARY:
The goal of this clinical trial is to compare the safety and accuracy of single-plane and real-time biplane ultrasound imaging in guiding hip joint injections and explore the application effects of imaging technology in hip joint injections.

DETAILED DESCRIPTION:
Real-time biplane imaging, an emerging ultrasound technology, uses a three-dimensional (3D) matrix transducer to display simultaneously he longitudinal and transverse intersecting planes on a single screen without requiring rotation of the transducer. The modality displays the puncture path in real-time and exhibits the spatial relationship between the needle tip and the target site, as well as surrounding structures during guided puncture. This technology significantly improves the puncture success rate and reduces complication rates in procedures such as the placement of intrahepatic bile duct drains and central venous catheters. However, this technology has not yet been implemented for hip joint injections. Therefore, we compared the safety and accuracy of single-plane and real-time biplane ultrasound imaging in guiding hip joint injections and explored the application effects of imaging technology in hip joint injections.

ELIGIBILITY:
Inclusion Criteria:

1.15 to 80 years of age; 2.hip joint pain and/or limited hip joint mobility; 3.physical examination and imaging studies indicating hip joint pathology; 4.pain duration exceeding 6 months with no significant improvement after conservative treatment; 5.patients scheduled for hip arthroscopy.

Exclusion Criteria:

1. a history of hip joint surgery;
2. the presence of lumbar disease, ankylosing spondylitis, or sacroiliac-joint pathology;
3. femoral head necrosis;
4. drug allergies;
5. inability to cooperate, or other contraindications to puncture.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The first-attempt success rate | during operation
  The proportion of successful entries into the anterior synovial recess and completion of medication injection on the first needle insertion, without adjusting needle tip direction
The final success rate | during operation
  The proportion of successful medication injections completed with no more than two needle insertions

SECONDARY OUTCOMES:
Puncture time | during operation
  The duration from the insertion of the puncture needle into the skin until saline can be injected into the joint cavity without significant resistance
The number of needle adjustments | during operation
  The number of times the puncture needle was retracted slightly and the insertion direction was adjusted upon noticing that the needle tip had deviated from the intended trajectory
The operator confidence score | during operation
  Based on the operator's level of confidence during the puncture process, with 1 point indicating a lack of confidence in the success of the first attempt, 2 points indicating moderate confidence, and 3 points indicating strong confidence
Complications | during operation
  Refer to adverse reactions occurring during the puncture process, including hematomas resulting from damage to surrounding blood vessels, pain or numbness due to nerve injury, toxic reactions caused by anesthetic entering the bloodstream, and postoperative infections

CONTACTS AND LOCATIONS:
Overall Officials: Mingbo Zhang, Study Chair — Chinese PLA General Hospital; Guozheng Zhao, Study Director — Chinese PLA General Hospital
Locations (1):
- The First Medical Center of the PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No